CLINICAL TRIAL: NCT01242345
Title: Clinical Value of Advanced Patient Monitoring With Capnography and Analysis of the Integrated Pulmonary Index During Interventional Upper Gastrointestinale Endoscopy
Brief Title: Capnography During Upper GI Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, Capnography During Upper GI Endoscopy, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Capno-Interventional 2011
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Capnography as an Adjunct to Standard Monitoring During Midazolam and Propofol Sedation for Interventional Upper GI Endoscopy
Keywords: Hypoxemia; Capnography; Integrated pulmonary index; Sedation; Propofol; Safety
MeSH Terms: conditions — Hypoxia | interventions — Capnography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention (No Intervention): Standard monitoring.
- Capnography (Experimental): Arm with capnographic monitoring
  Interventions: Device: Capnography

INTERVENTIONS:
Device: Capnography — Monitoring of the capnography curve for early detection of apnea
  Arms: Capnography

SUMMARY:
In this randomized controlled trial the utility of capnography and IPI gets evaluated. Hypoxemia may occur during sedation with midazolam and propofol. Whether hypoxemia may be prevented by an additional capnographic monitoring is subject of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Scheduled for interventional upper GI endoscopy with midazolam and propofol sedation

Exclusion Criteria:

* No informed consent
* ASA IV or V
* Emergency endoscopy
* Preexisting hypotension, bradycardia or hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | From the start to the end of endoscopy, i.e. from 0 h to approximately 2 h

SECONDARY OUTCOMES:
Further complications | From the start to the end of endoscopy, i.e. from 0 h to approximately 2 h

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Ruhr Universität Bochum, Bochum
  - Technische Universität München, München
  - Deutsche Klinik für Diagnostik, Wiesbaden

REFERENCES:
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079